CLINICAL TRIAL: NCT07059208
Title: Atrioventricular Nodal Ablation Versus Pulmonary Vein Isolation - Patient Centred Decisions
Acronym: AVENUE PACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunshine Coast Hospital and Health Service (Other)
Responsible Party: Principal Investigator, Matthew Tung, Principal Investigator, Sunshine Coast Hospital and Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVENUE PACE
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation ablation; Pulmonary vein isolation; Physiological pacing; atrioventricular nodal ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation (Active Comparator): Patients randomised to this arm would undergo catheter ablation targeted at achieving pulmonary vein isolation
  Interventions: Procedure: Pulmonary vein isolation
- Pacemaker implant and atrioventricular nodal ablation (Active Comparator): Patients randomised to this arm would undergo physiological pacing followed by atrioventricular nodal ablation
  Interventions: Procedure: Atrioventricular nodal ablation

INTERVENTIONS:
Procedure: Atrioventricular nodal ablation — Patients randomised to this arm would undergo physiological pacing followed by atrioventricular nodal ablation
  Arms: Pacemaker implant and atrioventricular nodal ablation
Procedure: Pulmonary vein isolation — Patients randomised to this arm would undergo catheter ablation targeted at achieving pulmonary vein isolation
  Arms: Pulmonary vein isolation

SUMMARY:
The goal of this clinical trial is to compare two procedural approaches to managing atrial fibrillation. The main questions it aims to answer are:

Is AF ablation or pacemaker implant and AV nodal ablation a more effective treatment approach for patients with atrial fibrillation refractory to pharmacological treatment?

What effect do these differing treatment approaches have on patient's quality of life and mental health?

Participants will:

Be randomly allocated to one of the treatment approaches. Visit the clinic 2 months, 12 months and 24 months after their procedure for a checkup, questionnaires and repeat heart ultrasounds.

DETAILED DESCRIPTION:
The goal of this trial is to compare the effectiveness and safety of pulmonary vein isolation compared with pacemaker implant and atrioventricular nodal ablation for patients with atrial fibrillation.

Patients who have been refractory to attempts at symptom control with pharmacological therapy will be eligible and will be randomised to one of the two approaches.

The primary outcome will be all cause rehospitalisation with secondary outcomes including procedural complications, echocardiographic measurements, patient reported outcomes, all cause mortality and rehospitalisation due to cardiovascular causes. These will be assessed over the 2 years following the index procedure.

The patient reported outcome measures will be the EQ5D, AF Effect on Quality of life score (AFEQT), Hospital anxiety and depression score (HADS) and Somatosensory amplification scale.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 65 years for patients with persistent atrial fibrillation or greater than 75 years for patients with paroxysmal atrial fibrillation.
* Unsuccessful trial of at least one pharmacological rate or rhythm control medication. This includes patients with medication refractory AF and/or intolerance to the medication(s).
* A resting ECG demonstrating AF with ventricular response rate >70bpm on a pharmacological rate control medication, or >90bpm while not on rate control medication.

Exclusion Criteria:

* Previous pulmomary vein isolation, left atrial flutter ablation or atrioventricular node ablation.
* BMI >40.
* Not suitable for pulmonary vein isolation and/or pacemaker implant on clinical grounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
All cause rehospitalisation | 2 years
  All rehospitalisations for any reason will be included

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data will be shared with any potential research collaborators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 Oct 2025 to 1 Oct 2035
Access Criteria: Accessible by contact person listed